CLINICAL TRIAL: NCT07265700
Title: Monocentric Prospective, Randomized, Non-blinded, Active-controlled Trial to Evaluate the Non-inferiority of Functional Magnetic Stimulation (FMS) on the Tesla Chair Compared to Physiotherapy in First or Second-degree Urinary Incontinence
Brief Title: Is Treatment With FMS Tesla Chair Equal to Physiotherapy in First and Second-degree Urinary Incontinence?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tesla-UI
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tesla-Chair (Experimental)
  Interventions: Device: Tesla-Chair
- Pelvicfloor physiotherapy (Active Comparator)
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Device: Tesla-Chair — Magnetic stimulation using the Tesla-Chair
  Arms: Tesla-Chair
Procedure: Physiotherapy — Pelvicfloor physiotherapy
  Arms: Pelvicfloor physiotherapy

SUMMARY:
100 patients with mild to moderate urinary incontinence will be randomly divided into two groups. One half will receive functional magnetic stimulation with the Tesla Chair for three months, while the other half will be treated with pelvic floor physiotherapy for the same period. After three and six months, a comparison will be made to determine which patient groups experience an improvement in urinary incontinence and how their muscle strength improves.

DETAILED DESCRIPTION:
Urinary incontinence is a debilitating condition that significantly impacts patients' quality of life, contributing to anxiety, depression, and social withdrawal. The severity of stress urinary incontinence (SUI) is directly correlated with increased physical and psychological burden. Although lifestyle modifications can offer moderate symptom relief, the current gold-standard first-line treatment is pelvic floor physiotherapy, with surgical intervention reserved for refractory cases.

Functional magnetic stimulation (FMS) has demonstrated positive effects in patients with urinary incontinence, including improvements in urodynamic parameters. However, limited research has directly compared the efficacy of FMS as a first-line therapy with standard pelvic floor physiotherapy. Addressing this gap is essential for informing clinical practice and expanding evidence-based therapeutic options. The efficacy of pelvic floor physiotherapy is commonly evaluated using the Oxford Scale, which provides an objective measure of pelvic floor muscle contraction strength. Additionally, patient-reported outcomes are assessed using validated instruments, including the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF UI) and the German Pelvic Floor Questionnaire (Deutscher Beckenbodenfragebogen), capturing symptom severity and quality of life. Together, these endpoints-objective assessments and patient-reported outcomes-offer a comprehensive evaluation of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Urinary incontinence of first or second degree
* Written informed consent
* German speaking (Study information and IC available only in German)

Exclusion Criteria:

* Pregnancy or desire to become pregnant
* Urinary incontinence of third degree
* Third or fourth degree pelvic organ prolapses
* no noticeable voluntary muscle activity according to Oxford = O/5
* Genital infections
* Malignant tumors
* Severe neurological diseases
* Cardiac arrhythmia
* Active internal medical devices e.g. cardiac pacemakers, medication pumps etc.
* Ferromagnetic implants at or near the site of stimulation
* Recent surgery at the site of stimulation
* Thrombosis or thrombophlebitis
* Epilepsy or suspected epilepsy
* Acute stages of kidney stones
* Gastrointestinal and internal disease at the site of stimulation
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* Previous enrolment into the current investigation
* Enrolment of the Sponsor or PI, their family members, employees and other dependent persons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in ICIQ-SF UI Score | 3 months post-treatment (6 months from baseline)
  Change in the International Consultation on Incontinence Questionnaire - Short Form for Urinary Incontinence (ICIQ-SF UI) score from baseline to 3 months after treatment; 1-5= slight incontinence, 19-21= very severe incontinence
Change in ICIQ-SF UI Score | 6-months post-treatment (9 months from baseline)
  Change in the International Consultation on Incontinence Questionnaire - Short Form for Urinary Incontinence (ICIQ-SF UI) score from baseline to 6 months after treatment

SECONDARY OUTCOMES:
Change in pelvic floor muscle strength, measured by the Oxford Scale | 3 months post-treatment (6 months from baseline)
  Change in pelvic floor muscle strength, measured by the Oxford Scale, 0= no contraction, 5= movement against gravity with full resistance.
Change in pelvic floor muscle strength, measured by the Oxford Scale | 6 months post-treatment (9 months from baseline)
  Change in pelvic floor muscle strength, measured by the Oxford Scale, 0= no contraction, 5= movement against gravity with full resistance.

IPD SHARING:
Plan to Share IPD: No